CLINICAL TRIAL: NCT00718211
Title: A Retrospective Clinical Records Review of Patients Diagnosed With Gastrointestinal Stromal Tumour at Two Tertiary Institutes in Singapore.
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: GA01/12/06
Record Dates: First submitted 2008-07-15; First posted 2008-07-18 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2014-01

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

SUMMARY:
To review the characteristics and treatment of gastrointestinal tumours at the two tertiary centres in Singapore

DETAILED DESCRIPTION:
A retrospective clinical records review of patients diagnosed with gastrointestinal stromal tumour (GIST) in the two tertiary centres in Singapore i.e. Singapore General Hospital and National University Hospital.

Gastrointestinal tumours are the most common soft-tissue tumours of the gastrointestinal tracts. Remarkable progress has been made during the last several years in the diagnosis and treatment of GIST. Understanding of the molecular pathogenesis of GIST which is linked to deregulated KIT tyrosine-kinase activity has improved diagnosis, such that GIST is now more frequently and specifically identified. More importantly, systemic tyrosine kinase inhibitor, imatinib, has been used successfully in the treatment of GIST patients with advanced or unresectable disease.

GIST has been reviewed in the Western literature but there is a lack of Asian data. The review will help us to better understand the disease in our population.Furthermore we will also examine several unresolved issues in the Western literature by looking into our local data. These include required duration of imatinib therapy, role of imatinib in the adjuvant setting (application of chemotherapy after macroscopically complete removal of tumour) and role of combination therapies.

The medical records of all patients diagnosed with the disease at the two centres will be reviewed.

Analysis of the results aims to:

1. to compare the characteristics of the GIST (epidemiology, site, morphology, immunohistochemistry profile) in our centres compared to the well-published literature.
2. to compare the treatment regimen and results of our centres compared to others
3. to review the role of chemotherapy in the adjuvant settings in the centres.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Gastrointestinal stromal tumor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: To review medical records of all patients diagnosed with the disease at the two specified centres.
  The medical records will be obtained through both paper and electronic medical systems.
  All data will be contained in a password secured database and will be securely located behind institutional firewalls.
Sampling Method: Probability Sample
Dates: Start 2006-05; Primary Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross Andrew Soo, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore